CLINICAL TRIAL: NCT05500014
Title: Effect of Altitude on Iron Absorption in Iron Depleted Women
Acronym: PotatoAlt
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Distance University of Applied Sciences (Other)
Collaborators: ETH Zurich (Switzerland) (Other); Instituto de Investigacion Nutricional, Peru (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022/01
Record Dates: First submitted 2022-07-11; First posted 2022-08-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Iron Deficiency Anemia; Iron Deficiency (Without Anemia); Altitude Hypoxia
Keywords: iron absorption; iron status; iron biofortification; Altitude and iron metabolism
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biofortified potato (Experimental): 500 g of biofortified, cooked potato, comsumed over 5 consecutive days (500g for each day, for a total of 2500 g of cooked potato). Potato meals will be labelled with a total of 3 mg 57FeSO4.
  Interventions: Other: Biofortified potato, not genetically modified

INTERVENTIONS:
Other: Biofortified potato, not genetically modified — Cooked potato, not genetically modified, with the addition of an acqueous solution of 57FeSO4 (3 mg in total).
  Other Names: Potato test meals

SUMMARY:
One of the most common nutritional deficiencies worldwide is iron deficiency. Iron deficiency is considered the main cause of anaemia in developing countries, including those in South America. The most recent surveys report that the prevalence of anaemia is as high as, 40 and 25% in Peru.

Populations living at higher altitudes may have higher iron requirements, as body iron is naturally increased in long-term high-altitude residents to compensate for the lower oxygen in the air at high altitudes. However, the effects of chronic exposure to high altitude on iron status, body iron compartments and dietary iron requirements are incompletely understood.

The primary objective of the proposed research is to determine iron bioavailability of iron from biofortified potatoes at different altitudes in populations of Andean descent. Human trials will be undertaken with volunteers in the Huancavelica region of Peru (elevation: 3676 meters) as well as in Lima (elevation close to sea level). The aim is to assess the effect of altitude on the absorption from a promising iron biofortified potato cultivar. These trials require incorporation of iron stable isotopes into the meals of the bio fortified potato and the analysis of the isotopes in subsequent blood (red blood cells) samples. Stable iron istotopes are considered the golden standard to assess human iron absorption and can be safely used as tracer substances in humans.

The objective of the study is to compare, in volunteer females of childbearing age, the bioavailability of iron from bio-fortified potatoes in two locations of different altitudes and quantify the effect of altitude on iron bioavailability from a potato meal consumed over 5 consecutive days.

DETAILED DESCRIPTION:
Populations living at higher altitudes may have higher iron requirements, as body iron is naturally increased in long-term high-altitude residents to compensate for the lower oxygen partial pressure. A residence altitude of 3600 masl implies an increase in Hemoglobin of ≈30 g Hb/l, which would correspond, in a 60 Kg woman to an increase of ≈500 mg red blood cell iron. Early studies in Bolivia have suggested decreased iron stores in women living at altitudes >3000 masl, compared to their counterparty living below 3000 masl .

The short-term exposure to high altitudes has profound impacts on iron metabolism. The lower oxygen partial pressure increases the rate of red blood cell synthesis, which is reflected in decrease in iron status parameters such as serum iron, serum ferritin, and an increase in erythropoietin and erythroferrone which in turn downregulate hepcidin, the master regulator of systemic iron metabolism , affecting iron release from stores and dietary iron absorption . In addition, intracellular oxygen sensors, the prolyl hydrolases (PHD's), stabilize hypoxia inducible factors (HIF-1α and HIF2-α) critically controlling transcriptional regulators such as dimetal transporter-1 (DMT-1) responsible for apical iron absorption in enterocytes .

Early studies in Peru by Huff et al. showed marked short-term increases of serum iron incorporation in red blood cells in subjects native from Lima (sea level) during acclimatization at Morococha, at 4540 masl. The opposite was the case in Morococha natives during acclimatization in Lima, as they had a decreased rate of plasma iron transfer to red blood cells . Notably however, during the short duration of the study (10 days) no marked change in red cell volume, hemoglobin or red cell mass could be detected.

Despite these well-described biologic mechanisms and short-term effects on physiological markers of iron status, the effects of chronic exposure to high altitude on iron status, body iron compartments and dietary iron requirements are incompletely understood. Genetic factors as reflected by different ethnicities are considered to play a large role in altitude-induced adaptations in iron metabolism .

A recent large study (n=71798) conducted in young male and iron replete Swiss army conscripts suggests a steady increase in hemoglobin and ferritin with increasing altitude, an increase that was detectable with each 300 masl increase, starting with as low as 300 masl of altitude. The authors also suggested that in this population, serum ferritin rose with altitude, independently from the increase in hemoglobin , suggesting a separate biological mechanism driving iron stores with increasing altitude. This data contrasts with data from Bolivia in apparently healthy women of reproductive age, where body iron stores were decreased at altitudes >3000 masl , compared to women living at lower altitudes (<3000 masl), suggesting that at high altitude, iron availability may be a limiting factor for optimal iron stores and for anemia prevention. More research is therefore needed on the determinants of iron balance in function of altitude, namely the interplay between dietary iron absorption, iron status, and iron status markers.

The primary objective of the proposed research is to determine iron bioavailability of iron from biofortified potatoes at different altitudes in populations of Andean descent. Human trials will be undertaken with volunteers in the Huancavelica region of Peru (elevation: 3676 meters) as well as in Lima (elevation close to sea level). The aim is to assess the effect of altitude on the absorption from a promising iron biofortified potato cultivar. These trials require incorporation of iron stable isotopes into the meals of the bio fortified and the analysis of the isotopes in subsequent blood (red blood cells) samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18-40 years
* Able to understand study requirements and provide written informed consent.
* Huancavelica study site: having been a Huancavelica or Peruvian highlands resident in the last 5 years, with at least one parent being from Huancavelica
* Lima study site: having been a Lima resident in the last 5 years, with origins and at least one parent being from the Peruvian highlands (>3000 masl)
* Serum ferritin at screening < 30 microgram/L

Exclusion Criteria:

* Illness that affects the nutritional status or food intake: gastrointestinal or renal problems; self-reported metabolic disease based on prior diagnosis, or a prior screening questionnaire.
* Pregnancy (positive urine test).
* Currently breastfeeding.
* Allergy to any ingredients of the test meal.
* C-reactive protein >5mg/100ml (representing inflammation)
* Smoker (>1 cigarette per day)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Iron absorption | 3 weeks
  Iron absorption will be assessed by measuring the shift in the iron isotopic composition in red blood cells, 14 days after the last test meal administration. Iron absoroption will be expressed as percentage of the total dose administered in the test meals (%)

SECONDARY OUTCOMES:
Serum ferritin (SF) | 5 minutes (combined with other biochemical assessements)
  Is a proxy of iron stores will be measured in human serum at baseline and is expressed in micrograms /liter serum
soluble transferrin receptor (sTfR) | 5 minutes (combined with other biochemical assessements)
  is expressed as mg/L human serum and will be assessed baseline
C-Reactive Protein (CRP) | 5 minutes (combined with other biochemical assessements)
  is an inflammatory marker and will be assessed at baseline in human serum at baseline
alpha acid glycoprotein (AGP) | 5 minutes (combined with other biochemical assessements)
  Is an inflammatory marker and will be assessed at baseline in human serum at baseline

OTHER OUTCOMES:
Socioeconomic, diet and physical activity | 1 hour
  A questionnaire will be completed with the subjects to assess socioeconomic factors, dietary patterns and physical activity
Erytropoietin | 5 minutes (combined with other biochemical assessements)
  Is a marker of erytroid activity and will be measured in human serum at baseline
Erythroferrone | 5 minutes (combined with other biochemical assessements)
  Is a marker of erytroid activity and will be measured in human serum at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — Swiss Distance University of Applied Sciences; Maria-Reyna Liria, PhD, Study Director — Insituto Investigation Nutritional
Locations (2):
- Peru (2):
  - Instituto International Nutrition, Huancavelica
  - Insituto National de Nutrition, Lima

IPD SHARING:
Plan to Share IPD: Undecided